CLINICAL TRIAL: NCT05811585
Title: Post-Market Clinical Follow-up Study for ADEPT® in Laparoscopic Gynecologic Surgery
Brief Title: PMCF Study for ADEPT® in LaparoscopicGynecologic Surgery
Status: Completed | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU562080
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Adhesion
Keywords: laparoscopic gynecologic surgery; adhesion-related morbidities
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patient of a Laparoscopic Gynecologic Surgery: ADEPT administered intraperitoneally as a liquid, used for irrigation throughout the procedure and for final instillation of a suitable amount at the end of the procedure.
  Interventions: Device: ADEPT

INTERVENTIONS:
Device: ADEPT — Adhesion Reduction Solution (4% icodextrin solution)

SUMMARY:
Postoperative adhesions develop in most patients after gynecologic surgery, likely resulting in significant morbidity, complications, and considerable increases in healthcare costs. Good surgical techniques, including a minimally invasive approach, may reduce adhesions and minimize the abovementioned complications. The agents for prevention or reduction of adhesion formation are placed inside the abdominal cavity, and especially in the pelvic cavity, which contains the female reproductive organs. ADEPT Adhesion Reduction Solution, hereinafter referred to as ADEPT, is intended for use as an intraperitoneal instillate for the reduction of adhesions following gynecological laparoscopic surgeries. The objective of this study is to evaluate the effectiveness and safety of ADEPT by detecting the incidence of adhesion-related morbidities (adhesion-related readmissions, including reoperations) after laparoscopic gynecologic surgery through a single-arm, retrospective, chart review with a patient questionnaire intended to supplement the patient chart.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients who, at the time of surgery, were ≥ 18 years of age and who had undergone an index laparoscopic gynecologic surgery at least 2 years prior to the start of the study.
* Patients in whom ADEPT® was used as an irrigant during the index laparoscopic gynecologic surgical procedure and as an intraperitoneal instillate for the reduction of adhesions following laparoscopic surgery.

Exclusion Criteria:

* Patients who had frank infection in the abdominopelvic cavity at the time of the surgery.
* Patients who were pregnant or nursing at the time of the surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of patients who underwent an index laparoscopic gynecologic surgery (performed at least 2 years prior to the start of the study) during which ADEPT (4% icodextrin solution) was used as an irrigant during the index laparoscopic gynecologic surgical procedure and as an intraperitoneal instillate for the reduction of adhesions.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hospital readmissions directly or possibly related to adhesions | Within 2 years of surgery
  Patient charts will be reviewed to collect data on readmissions related to adhesions, which are defined as:
  * Directly related to adhesions (adhesiolysis, non-operative readmissions for adhesions, and adhesiolysis operations on female reproductive tract);
  * Possibly related to adhesions (gynecological operations, abdominal surgery, and non-operative readmissions);
  * Open or laparoscopic reoperations that could potentially be complicated by present adhesions.

CONTACTS AND LOCATIONS:
Locations (2):
- Texas Fertility Center, Austin, Texas, United States
- Pius Hospital Oldenburg, Oldenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy